CLINICAL TRIAL: NCT07359547
Title: Minimally Invasive Bleb-Forming Surgical Approaches for Treating Primary Open-Angle Glaucoma: A Randomized Controlled Trial Comparing XEN®-63 Gel Stent and PRESERFLO® MicroShunt
Brief Title: Comparing XEN®-63 Gel Stent and PRESERFLO® MicroShunt
Acronym: MINI-BATTLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University Hospital, Bonn (Other); Hospital de Santa Maria, Lisbon (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S70640
Record Dates: First submitted 2026-01-12; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: GLAUCOMA 1, OPEN ANGLE, D (Disorder)
Keywords: Glaucoma; MIBS; Minimally Invasive Bleb-Forming Surgery; Bleb-Forming Devices Without a Plate; Surgery; PRESERFLO; MicroShunt; XEN; Gelstent
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRESERFLO MicroShunt (Experimental): The PFMS is a SIBS-polymer microshunt.
  Interventions: Device: PRESERFLO™ MicroShunt
- XEN 63 Gelstent (Active Comparator): The XEN 63 Gelstent is a hydrophilic gel implant made of cross-linked, purified collagen (gelatin).
  Interventions: Device: XEN®-63 Gel Stent

INTERVENTIONS:
Device: XEN®-63 Gel Stent — The XEN®-63 Gel Stent is a hydrophilic gel implant made of cross-linked, purified collagen (gelatin). This devices bypasses the trabecular meshwork and lower eye pressure via a subconjunctival filtering bleb, aided by intra-operative mitomycin C to reduce scarring. It has already been approved for the European market and therefore bear the CE mark.
  Arms: XEN 63 Gelstent
Device: PRESERFLO™ MicroShunt — The PRESERFLO™ MicroShunt is a SIBS-polymer microshunt. This devices bypasses the trabecular meshwork and lower eye pressure via a subconjunctival filtering bleb, aided by intra-operative mitomycin C to reduce scarring. It has already been approved for the European market and therefore bear the CE mark.
  Arms: PRESERFLO MicroShunt

SUMMARY:
The goal of this randomized controlled clinical trial is to learn whether two minimally invasive bleb-forming glaucoma implants can effectively treat adult patients with open-angle glaucoma who require surgical lowering of intraocular pressure (IOP). Specifically, the study evaluates whether the PRESERFLO™ MicroShunt is at least as effective as the XEN®-63 Gel Stent in reducing IOP after surgery. ￼

The main questions it aims to answer are:

* Does the PRESERFLO™ MicroShunt provide IOP reduction at 12 months that is non-inferior to the XEN®-63 Gel Stent?
* How do the two devices compare over 24 months with respect to medication reduction, need for additional glaucoma procedures, complications, and preservation of visual function and ocular structures?

Participants will:

* Be randomly assigned (1:1) to receive either the XEN®-63 Gel Stent or the PRESERFLO™ MicroShunt during a single glaucoma surgery.
* Attend scheduled follow-up visits over 24 months for eye-pressure measurements, vision testing, visual-field testing, OCT imaging, endothelial-cell counts, and safety assessments.
* Receive standard postoperative care and report any complications or additional treatments during the study period.

ELIGIBILITY:
Inclusion Criteria:

* >40 years of age
* An established diagnosis of: Primary open angle glaucoma, Normal tension glaucoma, Pigment dispersion glaucoma (PDG) or Pseudoexfoliative glaucoma (PEX)
* Inadequately controlled on maximum tolerated medical therapy.
* Mean Deviation (MD) </= -3
* Intraocular pressure of 14-28 mmHg
* Endothelial Cell Count ≥1000 cells/mm2

Exclusion Criteria:

* An established diagnosis of: Closed-angle glaucoma or Secondary open-angle glaucoma (besides PDG and PEX)
* Lens status: Aphakic patients or Anterior chamber intraocular lens
* Previous procedures: Glaucoma shunt/valve/ surgery or cyclodestructive procedure, Selective laser trabeculoplasty within the past 3 months, Incisional ophthalmic surgery involving the conjunctiva within the past 3 months, Clear corneal cataract or trabecular meshwork surgery conducted within the past 6 months.
* Presence of intraocular silicone oil
* No light perception vision
* Current corticosteroid use (ocular or oral)
* Conjunctival pathologies (e.g., pterygium)
* Active inflammation (e.g., blepharitis, conjunctivitis, keratitis, uveitis)
* Vitreous present in the anterior chamber
* Active iris neovascularization or neovascularization of the iris within 6 months of the surgical date
* Unwillingness or inability to give consent, accept randomization or return for and participate in scheduled protocol visits

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | 1 year

SECONDARY OUTCOMES:
Number of medications | 2 year
  Number of topical glaucoma medications
adverse events | 2 years
secundary pressure-lowering surgery | 2 years
Mean Deviation changes on the visual field | 2 years
Retinal Nerve Fibre Layer Thickness changes on Optical Coherence Tomography | 2 years
Endothelial Cell Count | 2 years
Best Corrected Visual Acuity | 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- University Hospitals UZ Leuven, Leuven, Vlaams-brabant, Belgium
- Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia, Germany
- ULS Santa Maria, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided